CLINICAL TRIAL: NCT04656249
Title: The Efficacy and Safety of Lenvatinib in Patients With Previously Treated Advanced Biliary Tract Cancer
Brief Title: Lenvatinib in Patients With Previously Treated Advanced Biliary Tract Cancer
Acronym: LENABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-JS-1391
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2020-11

CONDITIONS: Cholangiocarcinoma; Biliary Tract Cancer; Targeted Therapy
Keywords: Lenvatinib; Refractory biliary tract carcinoma; Efficacy; Biomarker
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: Patients are confirmed with biliary tract cancers by imaging and histological examination and meet with the inclusive criteria, including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, common bile duct cancer and gallbladder cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib (Experimental): Drug doses for BTC are identical, being orally administered at 8mg/d to patients weighing <60 kg and 12mg/d to those ≥60 kg.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Drug doses for BTC are identical, being orally administered at 8mg/d to patients weighing <60 kg and 12mg/d to those ≥60 kg.
  Other Names: E7080; Lenvima

SUMMARY:
This is a single center, nonrandom, open-label study aiming to evluate the efficacy and safety of lenvatinib for patients with pretreated advanced biliary tract cancer.

DETAILED DESCRIPTION:
Lenvatinib targets VEGFR1, 2, and 3, PDGFRα, Fibroblast growth factor receptor (FGFR), and the KIT and RET tyrosine kinases and was initially developed for use in various tumor types. This is a single-center, non-random, open-label study in participants with unresectable BTC and disease progression or failure following at least one chemotherapy regimen. This study contains three procedures: a pre-treatment procedure that will last within 21 days; a treatment procedure that will consist of study treatment cycles and tumor assessment conducted every 6-8 weeks; and a follow-up procedure that will begin immediately after the off-treatment visit and will continue as long as the participant is alive, unless the participant withdraws consent, or until the terminal of the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Pathologically or cytologically confirmed adenocarcinoma of biliary tract cancer (intrahepatic, extrahepatic cholangiocarcinoma, gall bladder cancer), at least one prior chemotherapy.
  2. Participants who received adjuvant chemotherapy are eligible if this therapy was completed and recurrent has not been shown for 6 months after the completion of the therapy
  3. Measurable disease meeting the following criteria: At least 1 lesion of ≥ 1.0 cm in the longest diameter for a non-lymph node or ≥ 1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1) using computerized tomography/magnetic resonance imaging (CT/MRI). Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
  4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
  5. Survival expectation of 3 months or longer after beginning of study treatment
  6. Males or females age ≥ 18 years at the time of informed consent
  7. All chemotherapy- or radiation-related toxicities must have resolved to Grade 0-1 per Common Terminology Criteria for Adverse Events (CTCAE v 4.03), except alopecia, infertility, and the adverse events listed in inclusion criteria
  8. Adequately controlled blood pressure (BP) with or without antihypertensive medications (defined as BP ≤ 150/90 mm Hg at Screening and no change in antihypertensive medications within 1 week prior to the first dose of study drug)
  9. Participants with adequate function of major organs and blood coagulation:
  10. Absolute neutrophil count (ANC) ≥ 1500/mm^3 ( ≥ 1.5×103/μl); Platelets ≥ 100,000/mm3 ( ≥ 100×10^9/L); Hemoglobin ≥ 9.0 g/dL; Bilirubin ≤ 2.0 mg/dL except for unconjugated hyperbilirubinemia or Gilbert's syndrome; Alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN) ( ≤ 5.0 × ULN for participants with the liver metastasis); Creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula; Prothrombin time-International Normalized Ratio (PT-INR) ≤ 1.5;
  11. Participants must voluntarily agree to provide written informed consent;
  12. Participants must be willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Ascites of moderate, severe, or requiring drainage
2. Proteinuria of ≥ 2+ on dipstick testing (Grade ≤ 1 confirmed by quantitative assessment is eligible)
3. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of study drug
4. New York Heart Association congestive heart failure of class II or above, unstable angina, myocardial infarction, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months from the first dose of study drug
5. A prolonged QT/QTc interval (QTcF > 480 ms)
6. Known to be human immunodeficiency virus (HIV) positive
7. Active infection requiring systemic treatment
8. Bleeding or thrombotic disorders or chronic systemic use of anticoagulants requiring therapeutic INR monitoring, eg, warfarin or similar agents (treatment with low molecular weight heparin is permitted)
9. Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 21 days prior to the first dose of study drug Active malignancy (except for BTC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, carcinoma in-situ of the cervix, or early stage gastric/colorectal cancer) within the past 24 months prior to the first dose of study drug
10. Known intolerance to the study drug or any of the excipients
11. History of drug or alcohol dependency or abuse within the last 24 months prior to the first dose of study drug
12. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study
13. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive human chorionic gonadotropin [hCG or B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 3 days before the first dose of study drug.
14. For either males unless undergoing a successful vasectomy (confirmed azoospermia) or females of childbearing potential, the participant and his/her partner do not agree to use a medically appropriate method of contraception throughout the entire study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Six months
  Objective response rate
Progression free survival (PFS) | Six months
  Progression free survival

SECONDARY OUTCOMES:
Overall survival (OS) | Two years
  Overall survival (OS) [ Time Frame: From the date of first dose of study drug to the date of death from any cause, or up to approximately 2 years ]
Disease control rate (DCR) | Six months
  DCR is defined as the percentage of participants with complete response (CR) + partial response (PR) + stable disease (SD).
The Rate of Treatment Related Adverse Events | Three years
  Treatment related adverse events (AEs) were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE 4.0). The study recorded the occurrence rate of treatment related AEs

OTHER OUTCOMES:
Clinical benefit rate (CBR) | One years
  Clinical benefit rate (CBR) [ Time Frame: From the date of first dose of study drug to the date of the first documentation of disease progression or death from any cause, whichever occurs first, or up to approximately 1 years ]

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Tao Zhao, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Result] Marquardt JU, Saborowski A, Czauderna C, Vogel A. The Changing Landscape of Systemic Treatment of Advanced Hepatocellular Carcinoma: New Targeted Agents and Immunotherapies. Target Oncol. 2019 Apr;14(2):115-123. doi: 10.1007/s11523-019-00624-w. PMID 30805831
- [Result] Obi S, Sato T, Sato S, Kanda M, Tokudome Y, Kojima Y, Suzuki Y, Hosoda K, Kawai T, Kondo Y, Isomura Y, Ohyama H, Nakagomi K, Ashizawa H, Miura Y, Amano H, Mochizuki H, Omata M. The efficacy and safety of lenvatinib for advanced hepatocellular carcinoma in a real-world setting. Hepatol Int. 2019 Mar;13(2):199-204. doi: 10.1007/s12072-019-09929-4. Epub 2019 Jan 22. PMID 30671808
- [Result] Hiraoka A, Kumada T, Kariyama K, Takaguchi K, Atsukawa M, Itobayashi E, Tsuji K, Tajiri K, Hirooka M, Shimada N, Shibata H, Ishikawa T, Ochi H, Tada T, Toyoda H, Nouso K, Tsutsui A, Itokawa N, Imai M, Joko K, Hiasa Y, Michitaka K; Real-life Practice Experts for HCC (RELPEC) Study Group, HCC 48 Group (hepatocellular carcinoma experts from 48 clinics in Japan). Clinical features of lenvatinib for unresectable hepatocellular carcinoma in real-world conditions: Multicenter analysis. Cancer Med. 2019 Jan;8(1):137-146. doi: 10.1002/cam4.1909. Epub 2018 Dec 21. PMID 30575325
- [Result] El-Serag HB. Epidemiology of viral hepatitis and hepatocellular carcinoma. Gastroenterology. 2012 May;142(6):1264-1273.e1. doi: 10.1053/j.gastro.2011.12.061. PMID 22537432
- [Result] Zhang B, Zhang B, Zhang Z, Huang Z, Chen Y, Chen M, Bie P, Peng B, Wu L, Wang Z, Li B, Fan J, Qin L, Chen P, Liu J, Tang Z, Niu J, Yin X, Li D, He S, Jiang B, Mao Y, Zhou W, Chen X. 42,573 cases of hepatectomy in China: a multicenter retrospective investigation. Sci China Life Sci. 2018 Jun;61(6):660-670. doi: 10.1007/s11427-017-9259-9. Epub 2018 Feb 2. PMID 29417360
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Witjes CD, Karim-Kos HE, Visser O, de Vries E, IJzermans JN, de Man RA, Coebergh JW, Verhoef C. Intrahepatic cholangiocarcinoma in a low endemic area: rising incidence and improved survival. HPB (Oxford). 2012 Nov;14(11):777-81. doi: 10.1111/j.1477-2574.2012.00536.x. Epub 2012 Aug 17. PMID 23043667
- [Result] Bridgewater J, Galle PR, Khan SA, Llovet JM, Park JW, Patel T, Pawlik TM, Gores GJ. Guidelines for the diagnosis and management of intrahepatic cholangiocarcinoma. J Hepatol. 2014 Jun;60(6):1268-89. doi: 10.1016/j.jhep.2014.01.021. Epub 2014 Mar 27. No abstract available. PMID 24681130
- [Result] Ueno M, Ikeda M, Sasaki T, Nagashima F, Mizuno N, Shimizu S, Ikezawa H, Hayata N, Nakajima R, Morizane C. Phase 2 study of lenvatinib monotherapy as second-line treatment in unresectable biliary tract cancer: primary analysis results. BMC Cancer. 2020 Nov 16;20(1):1105. doi: 10.1186/s12885-020-07365-4. PMID 33198671
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Zhou J, Sun HC, Wang Z, Cong WM, Wang JH, Zeng MS, Yang JM, Bie P, Liu LX, Wen TF, Han GH, Wang MQ, Liu RB, Lu LG, Ren ZG, Chen MS, Zeng ZC, Liang P, Liang CH, Chen M, Yan FH, Wang WP, Ji Y, Cheng WW, Dai CL, Jia WD, Li YM, Li YX, Liang J, Liu TS, Lv GY, Mao YL, Ren WX, Shi HC, Wang WT, Wang XY, Xing BC, Xu JM, Yang JY, Yang YF, Ye SL, Yin ZY, Zhang BH, Zhang SJ, Zhou WP, Zhu JY, Liu R, Shi YH, Xiao YS, Dai Z, Teng GJ, Cai JQ, Wang WL, Dong JH, Li Q, Shen F, Qin SK, Fan J. Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2017 Edition). Liver Cancer. 2018 Sep;7(3):235-260. doi: 10.1159/000488035. Epub 2018 Jun 14. PMID 30319983
- [Result] Ji X, Bu ZD, Yan Y, Li ZY, Wu AW, Zhang LH, Zhang J, Wu XJ, Zong XL, Li SX, Shan F, Jia ZY, Ji JF. The 8th edition of the American Joint Committee on Cancer tumor-node-metastasis staging system for gastric cancer is superior to the 7th edition: results from a Chinese mono-institutional study of 1663 patients. Gastric Cancer. 2018 Jul;21(4):643-652. doi: 10.1007/s10120-017-0779-5. Epub 2017 Nov 22. PMID 29168120
- [Result] Al-Salama ZT, Syed YY, Scott LJ. Lenvatinib: A Review in Hepatocellular Carcinoma. Drugs. 2019 Apr;79(6):665-674. doi: 10.1007/s40265-019-01116-x. PMID 30993651
- [Result] Zhu RX, Seto WK, Lai CL, Yuen MF. Epidemiology of Hepatocellular Carcinoma in the Asia-Pacific Region. Gut Liver. 2016 May 23;10(3):332-9. doi: 10.5009/gnl15257. PMID 27114433
- [Result] Ghidini M, Pizzo C, Botticelli A, Hahne JC, Passalacqua R, Tomasello G, Petrelli F. Biliary tract cancer: current challenges and future prospects. Cancer Manag Res. 2018 Dec 28;11:379-388. doi: 10.2147/CMAR.S157156. eCollection 2019. PMID 30643463
- [Result] Sohal DP, Mykulowycz K, Uehara T, Teitelbaum UR, Damjanov N, Giantonio BJ, Carberry M, Wissel P, Jacobs-Small M, O'Dwyer PJ, Sepulveda A, Sun W. A phase II trial of gemcitabine, irinotecan and panitumumab in advanced cholangiocarcinoma. Ann Oncol. 2013 Dec;24(12):3061-5. doi: 10.1093/annonc/mdt416. Epub 2013 Oct 20. PMID 24146220
- [Result] Snyder A, Morrissey MP, Hellmann MD. Use of Circulating Tumor DNA for Cancer Immunotherapy. Clin Cancer Res. 2019 Dec 1;25(23):6909-6915. doi: 10.1158/1078-0432.CCR-18-2688. Epub 2019 Jul 8. PMID 31285372
- [Result] Wang D, Lin J, Yang X, Long J, Bai Y, Yang X, Mao Y, Sang X, Seery S, Zhao H. Combination regimens with PD-1/PD-L1 immune checkpoint inhibitors for gastrointestinal malignancies. J Hematol Oncol. 2019 Apr 24;12(1):42. doi: 10.1186/s13045-019-0730-9. PMID 31014381
- [Result] Valle JW, Lamarca A, Goyal L, Barriuso J, Zhu AX. New Horizons for Precision Medicine in Biliary Tract Cancers. Cancer Discov. 2017 Sep;7(9):943-962. doi: 10.1158/2159-8290.CD-17-0245. Epub 2017 Aug 17. PMID 28818953
- [Result] Vokes EE, Ready N, Felip E, Horn L, Burgio MA, Antonia SJ, Aren Frontera O, Gettinger S, Holgado E, Spigel D, Waterhouse D, Domine M, Garassino M, Chow LQM, Blumenschein G Jr, Barlesi F, Coudert B, Gainor J, Arrieta O, Brahmer J, Butts C, Steins M, Geese WJ, Li A, Healey D, Crino L. Nivolumab versus docetaxel in previously treated advanced non-small-cell lung cancer (CheckMate 017 and CheckMate 057): 3-year update and outcomes in patients with liver metastases. Ann Oncol. 2018 Apr 1;29(4):959-965. doi: 10.1093/annonc/mdy041. PMID 29408986
- [Result] Matsuki M, Hoshi T, Yamamoto Y, Ikemori-Kawada M, Minoshima Y, Funahashi Y, Matsui J. Lenvatinib inhibits angiogenesis and tumor fibroblast growth factor signaling pathways in human hepatocellular carcinoma models. Cancer Med. 2018 Jun;7(6):2641-2653. doi: 10.1002/cam4.1517. Epub 2018 May 7. PMID 29733511